CLINICAL TRIAL: NCT00973726
Title: The Retinal Function in Relation to Glucose Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Stig Holfort, Glostrup Hospital, department of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Stig Holfort
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose Tolerance Test; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glucose (Other): Subjects are given an oral glucose tolerance test.
  Interventions: Other: Glucose test

INTERVENTIONS:
Other: Glucose test — Subjects ingest an oral glucose tolerance test.
  Other Names: Standardized oral glucose tolereance test (75 g glucose)

SUMMARY:
This project has the following specific purposes:

* To develop a clinically usable test to determine the blood glucose level or HbA1c-level, to which the retina is adapted. This will be performed by means of ERG implicit time measurements in relation to the blood glucose level during an oral glucose tolerance test (OGTT) and inter- or extrapolation to the level of blood glucose (or HbA1c) where implicit time is normal.
* To examine darkadaptation in diabetics in relation to changes in the glucose level.
* To examine vessel diameter changes in diabetic individuals when changing the glucose level transiently

DETAILED DESCRIPTION:
Study 1: 24 type 2 diabetics with minimal diabetic retinopathy but varying HbA1c level.

Study 2: 24 type 2 diabetics with minimal diabetic retinopathy. Study 3: 24 type 2 diabetics with minimal diabetic retinopathy.

Plan of trial:

Study 1: Test individuals will be examined at baseline: Prior history of illness, eye examination, blood test, fundusphoto and fullfield-ERG. Afterwards test individuals will take an oral glucose tolerance test (OGTT) which results in a peak in blood glucose after approx. 2 hours, whereafter the blood glucose level normalizes. Immediately after the sugar intake test individuals will be examined by repeated fullfield-ERG's and blood glucose measurements (every 30 min) until the blood glucose level has been normalized.

Study 2: Test individuals will be examined at baseline: Prior history of illness, eye examination, blood test, fundusphoto and dark adaptation. Afterwards test individuals will take an oral glucose tolerance test (OGTT) which results in a peak in blood glucose after approx. 2 hours, whereafter the blood glucose level normalizes. 80 minutes after the sugar intake test individuals will be examined by repeated dark adaptation and blood glucose measurements.

Study 3: Test individuals will be examined at baseline: Prior history of illness, eye examination, blood test, fundusphoto. Afterwards test individuals will take an oral glucose tolerance test (OGTT) which results in a peak in blood glucose after approx. 2 hours, whereafter the blood glucose level normalizes. At baseline (fasting) and 80 minutes after the sugar intake test individuals will be examined by redfree photos of optic disc and blood glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic individuals. Age > 17 < 80
* Dysregulated type 1 diabetic individuals and newly diagnosed type 1 diabetics. Age >17 < 60 years
* with minimal or no diabetic retinopathy defined by no more than five microaneurysms or dot hemorrhages per eye on three non-stereoscopic 50 degree color fundus photographs

Exclusion Criteria:

* Test individuals with significant cataract, prior surgery to the eye, diabetic retinopathy, other serious eye disease, hypertension, other serious systemic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Changes in amplitude/implicit times, changes in dark adaptation, changes in vessel caliber, changes in Optical coherence tomography (OCT) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stig Holfort, Medical Doctor, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark